CLINICAL TRIAL: NCT04445649
Title: Investigation of Prognostic Factors to Regain Consciousness in Neurological Early Rehabilitation
Brief Title: Prognostic Factors to Regain Consciousness
Status: Recruiting | Type: Observational
Sponsor: BDH-Klinik Hessisch Oldendorf (Other)
Responsible Party: Sponsor
Other Study IDs: DOC-OUT
Record Dates: First submitted 2020-06-18; First posted 2020-06-24 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Neurologic Disorder; Disorder of Consciousness; Traumatic Brain Injury; Stroke; Hypoxic-Ischemic Encephalopathy
Keywords: Neurological rehabilitation; Prognosis; Outcome; Level of consciousness
MeSH Terms: conditions — Nervous System Diseases; Consciousness Disorders; Brain Injuries, Traumatic; Stroke; Hypoxia-Ischemia, Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ICU patients: Patients with impaired consciousness admitted to intensive care unit after severe brain injury
  Interventions: Diagnostic Test: Coma-Recovery-Scale-Revised (CRS-R)

INTERVENTIONS:
Diagnostic Test: Coma-Recovery-Scale-Revised (CRS-R) — CRS-R assessments (15 minutes) are repeated weekly after study entry

SUMMARY:
The study aims to identify factors that predict the medium and long-term outcome of patients with disorders of consciousness (DOC) undergoing early neurological rehabilitation.

In this prospective, observational study, 130 DOC patients are going to be included (36 months). At study entry, different routine data, disease severity and functional status are documented for each patient. In addition, MRI, EEG and evoked potentials are measured within the first week. The level of consciousness is recorded with the Coma-Recovery-Scale-Revised and serves as the primary outcome parameter. Complications, comorbidities, functional status and leve of consciousness are assessed weekly. After eight weeks, the measurement of the MRI, the EEG and the evoked potentials are repeated. After 3, 6 and 12 months, the Glasgow Outcome Scale-Revised is used to followed up the current status of the patients.

DETAILED DESCRIPTION:
Due to continuous improvements in acute medical care, the number of patients surviving severe brain damage has increased over the past decades. While some patients improve significantly during the first days after the injury, other patients remain in altered states of consciousness (i.e. coma, unresponsive wakefulness syndrome or minimally conscious state). Acquired brain damage such as cerebrovascular diseases, traumatic brain injuries or hypoxic-ischemic encephalopathies are the main causes of severe impaired consciousness.The correct classification of the level of consciousness is of great importance, since the different states of consciousness are associated with different prognoses and treatment options. Patients who show minimal signs of consciousness (MCS) a month after the onset of the disease have better chances of regaining consciousness within one year than UWS patients. Within both categories (UWS, MCS), traumatic aetiologies in turn have a better prognosis than non-traumatic aetiologies. The prognosis usually begins with the admission of the patients to the intensive care unit of the acute care facility. But even in later treatment phases, a large number of patients regain consciousness, e.g. during post-acute early rehabilitation and even years after the disease. Numerous factors are associated with the prognosis (e.g. age, aetiology, duration of illness, functional status and state of consciousness). Although there are numerous studies on the prognostic factors and outcome of patients with severe brain damage, only a few have explicitly examined patients with initially severe and long-lasting impaired consciousness. The study therefore aims to identify factors that predict the medium and long-term outcome of patients with severe impaired consciousness in early neurological rehabilitation.

Over a period of 36 months, 130 patients undergoing neurological early rehabilitation with impaired consciousness are included. It is a prospective observational study that is carried out in a single neurological rehabilitation centre (monocentric). Different routine data, disease severity and functional status are documented for each patient. In addition, MRI, EEG and evoked potentials are measured within the first week. The level of consciousness is recorded with the Coma-Recovery-Scale-Revised and serves as the primary outcome parameter. Complications, comorbidities, functional status and leve of consciousness are assessed weekly. After eight weeks, the measurement of the MRI, the EEG and the evoked potentials are repeated. After 3, 6 and 12 months, the Glasgow Outcome Scale-Revised is used to follow up the current status of the patients.

ELIGIBILITY:
Inclusion Criteria:

* early neurological rehabilitation (phase B)
* stroke, traumatic brain injury, hypoxic-ischemic encephalopathy
* disorder of consciousness (coma, UWS, MCS)
* at minimum two weeks after disease onset
* admission to intensive care unit
* written consent from the patient's legal representative
* exclusion of pregnancy

Exclusion Criteria:

* insufficient cardiorespiratory stability
* fractures or severe infratentorial brain injuries leading to impaired auditory evoked - potentials
* previous brain damage
* mental disorders (dementia, depression)
* colonization with multi-resistant pathogens
* MRI contraindications
* claustrophobia
* weight > 120 kg

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing neurological early rehabilitation with impaired consciousness and admitted to intensive care unit
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Changed functional status | 8 weeks
  Functional status is measured with Early Rehabilitation Barthel Index (ERBI; Range: -325 to 100; higher scores mean a better outcome) weekly.

SECONDARY OUTCOMES:
Changed level of consciousness | 8 weeks
  Level of consciousness is measured with the Coma-Recovery-Scale-Revised (CRS-R; Range: 0 to 23; higher scores mean a better outcome) weekly.
Duration until consciousness is regained | up to 8 weeks
  Time until patients show first signs of consciousness

CONTACTS AND LOCATIONS:
Overall Officials: Jens D Rollnik, MD, Study Director — BDH-Clinic Hessisch Oldendorf; Melanie Boltzmann, PhD, Principal Investigator — BDH-Clinic Hessisch Oldendorf
Locations (1):
- BDH-Clinic Hessisch Oldendorf, Hessisch Oldendorf, Germany

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Period of availability begins when results are published, at the earliest in Dec 2023
Access Criteria: IPD can be obtained from the principal investigator upon reasonable request.

REFERENCES:
- [Background] Lucca LF, Lofaro D, Pignolo L, Leto E, Ursino M, Cortese MD, Conforti D, Tonin P, Cerasa A. Outcome prediction in disorders of consciousness: the role of coma recovery scale revised. BMC Neurol. 2019 Apr 18;19(1):68. doi: 10.1186/s12883-019-1293-7. PMID 30999877
- [Background] Portaccio E, Morrocchesi A, Romoli AM, Hakiki B, Taglioli MP, Lippi E, Di Renzone M, Grippo A, Macchi C; Intensive Rehabilitation Unit Study Group of the IRCCS Don Gnocchi Foundation, Italy. Improvement on the Coma Recovery Scale-Revised During the First Four Weeks of Hospital Stay Predicts Outcome at Discharge in Intensive Rehabilitation After Severe Brain Injury. Arch Phys Med Rehabil. 2018 May;99(5):914-919. doi: 10.1016/j.apmr.2018.01.015. Epub 2018 Feb 8. PMID 29428346
- [Background] Portaccio E, Morrocchesi A, Romoli AM, Hakiki B, Taglioli MP, Lippi E, Di Renzone M, Grippo A, Macchi C. Score on Coma Recovery Scale-Revised at admission predicts outcome at discharge in intensive rehabilitation after severe brain injury. Brain Inj. 2018;32(6):730-734. doi: 10.1080/02699052.2018.1440420. Epub 2018 Feb 26. PMID 29482376
- [Background] Estraneo A, Moretta P, Loreto V, Lanzillo B, Cozzolino A, Saltalamacchia A, Lullo F, Santoro L, Trojano L. Predictors of recovery of responsiveness in prolonged anoxic vegetative state. Neurology. 2013 Jan 29;80(5):464-70. doi: 10.1212/WNL.0b013e31827f0f31. Epub 2013 Jan 9. PMID 23303855
- [Background] Estraneo A, Moretta P, Loreto V, Lanzillo B, Santoro L, Trojano L. Late recovery after traumatic, anoxic, or hemorrhagic long-lasting vegetative state. Neurology. 2010 Jul 20;75(3):239-45. doi: 10.1212/WNL.0b013e3181e8e8cc. Epub 2010 Jun 16. PMID 20554941